CLINICAL TRIAL: NCT07129759
Title: A Long-term Extension Study to Evaluate the Safety and Tolerability of Daily Oral LUM-201 in Children With Growth Hormone Deficiency (GHD)
Brief Title: Phase 3 Long Term Safety Extension Study of LUM-201 in Children With Growth Hormone Deficiency
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-201-11
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Growth Hormone Deficiency (GHD)
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM-201 (Experimental)
  Interventions: Drug: LUM-201

INTERVENTIONS:
Drug: LUM-201 — 1.6 mg/kg/day, administered orally once daily

SUMMARY:
This is a Multi-national Trial. The Goal of the Trial is to Offer Subjects Who Complete 12 Months in the LUM-201-10 Phase 3 Trial up to an Additional 36 Months of Treatment of LUM-201 While Evaluating Safety and Tolerability of LUM-201.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver must be willing to provide written informed consent, and the subject must sign the assent, as applicable.
* Subject must have successfully completed 12 months of participation in the LUM-201 Phase 3 GHD trial, and be eligible for continuation of treatment, pending all other enrollment criteria are met.
* Subject who is sexually active must use an acceptable form of contraception.
* Subject must be eligible for the Day 1 visit as confirmed by the Investigator.

Exclusion Criteria:

* Subject has a medical or genetic condition that, in the opinion of the Investigator and/or MMs, adds unwarranted risk to use of LUM-201.
* Pregnancy.
* Subject has planned or is receiving current long-term treatment with medications known to prolong the QT interval or act as substrates, inducers, or inhibitors of the cytochrome system cytochrome P450 type 3A4 that metabolizes LUM-201 (see Appendix 6 for list of example medications). Subjects receiving shorter-term (two weeks or less) treatment with these medications should be evaluated on case-by-case basis by the Investigator in consultation with the MMs.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of LUM-201 | Day 1 - Month 36
  * The number of subjects with at least 1 (serious) treatment-related adverse event (TEAE).
  * The number of subjects with at least 1 suspected unexpected serious adverse reaction.
  * The number of subjects with clinically significant abnormalities related to trial laboratory tests or electrocardiograms (ECGs).
  * The number of subjects with at least 1 adverse event of special interest (AESI).
  * Annual change from baseline in body weight standard deviation score (SDS).
  * Annual change from baseline in body mass index (BMI) SDS.

SECONDARY OUTCOMES:
To evaluate the long-term effect of LUM-201 on growth. | Day 1 - Month 36
  * Annual height velocity.
  * Annual change in height standard deviation score (SDS).
  * Annual change in body mass index (BMI).
  * Annual change in BMI SDS.
  * Annual change in bone age (BA)/chronological age (CA) ratio.
To evaluate the long-term effect of LUM-201 on pharmacodynamic (PD) markers. | Day 1 - Month 36
  * Annual change in insulin-like growth factor (IGF)-1 SDS.
  * Annual change in insulin-like growth binding protein 3 (IGFBP-3) SDS.

IPD SHARING:
Plan to Share IPD: Undecided